CLINICAL TRIAL: NCT02158403
Title: PREVENtion of HeartMate II Pump Thrombosis Through Clinical Management
Brief Title: PREVENtion of HeartMate II Pump Thrombosis
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TC05232014
Record Dates: First submitted 2014-05-30; First posted 2014-06-06 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: HeartMate II Pump Thrombosis
Keywords: HeartMate II; heart assist device; pump thrombosis; hypercoagulable disorder; thrombus; Thoratec Corporation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinical Management Recommendations (Other): Clinical management recommendations for reducing pump thrombosis
  Interventions: Other: Clinical Management Recommendations for reducing pump thrombosis

INTERVENTIONS:
Other: Clinical Management Recommendations for reducing pump thrombosis — Clinical Management Recommendations for reducing pump thrombosis

SUMMARY:
The purpose of this study is to assess how often blood clots form in the FDA-approved HeartMate® II (HM II) Left Ventricular Assist Device (LVAD) and to identify risks related to clotting within the pump.

DETAILED DESCRIPTION:
PREVENT is a prospective, multi-center, non-randomized study that is designed (1) to assess the incidence of HM II pump thrombosis in the current era when recommended practices for clinical management are adopted, and (2) to identify the risk factors associated with pump thrombosis events. The recommended practices are focused on implantation technique, anticoagulation regimen, pump speed and blood pressure management. All consecutive patients receiving a HM II implant will be considered for this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative has signed an informed consent form
* Subject is receiving the HeartMate II as their first Left Ventricular Assist Device (LVAD)

Exclusion Criteria:

* Prior mechanical circulatory support (MCS) (except for intra-aortic balloon pump)
* Participation in any other clinical investigation(s) involving a MCS device, or an investigation(s) that is likely to confound study results or affect study outcome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of confirmed pump thrombosis within three months of HeartMate II (HM II) implantation | 3 months

SECONDARY OUTCOMES:
Incidence of confirmed pump thrombosis within six months of HM II implantation | 6 months
Incidence of suspected pump thrombosis (including unexplained hemolysis) within three and six months of HM II implantation | 3 and 6 months
Incidence of pump exchange, urgent transplantation or death due to pump thrombosis within three and six months of HM II implantation | 3 and 6 months
Survival on LVAD support at six months post HM II implantation | 6 months
Multivariate analysis of risk factors for pump thrombosis including demographics, anti-coagulation regimen, selected laboratory data (INR, LDH, plasma free Hgb), pump position measures, pump parameters and blood pressure | Baseline and 1 week, 1 month, 3 months and 6 months after surgery
Subgroup analysis of subjects identified as having a hypercoagulable disorder prior to HM II implantation | Baseline and 3 months after implant
Characterization of pump position in the study population (measured via quantitative assessment of X-ray images including inflow cannula angle, outflow cannula angle and pump pocket depth) | 1 week and 6 months after surgery
Characterization of selected lab values (INR, LDH and plasma free Hgb) within the study population | Baseline, 1 week (plus or minus 3 days), 1 month (plus or minus 7 days), 3 months and 6 months (plus or minus 30 days) after surgery
Incidence of protocol-defined anticipated adverse events | Baseline, 1 month , 3 months and 6 months after surgery
Characterization of pump parameters in the study population including power (watts), speed (rpm), flow (L/min), and pulsatility index | 1 week, 1 month, 3 months, and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Sundareswaran, PhD, Study Director — Abbott
Locations (23):
- United States (23):
  - Baptist Medical Center, Little Rock, Arkansas
  - University of California, San Diego, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Sutter Memorial, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Shands Hospital at University of Florida, Gainesville, Florida
  - Northwestern Memorial, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Jewish Hospital, Louisville, Kentucky
  - Abbott Northwestern, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, St. Mary's, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Memorial Hermann/UT Texas, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- [Derived] Jeske W, Ransom J, Katz JN, Kilic A, Lindenfeld J, Egnaczyk G, Shah P, Brieke A, Uriel N, Crandall D, Farrar DJ, Walenga JM. Enhanced Thrombin Formation in Patients With Ventricular Assist Devices Experiencing Bleeding: Insights From the Multicenter PREVENT Study. ASAIO J. 2023 Mar 1;69(3):278-283. doi: 10.1097/MAT.0000000000001790. Epub 2022 Sep 8. PMID 36731068
- [Derived] Kilic A, Ransom J, Maltais S, Sun B, Entwistle JW 3rd, Bailey S, John R, Klodell CT, Gregoric I, Sheridan B, Chuang J, Farrar DJ, Sundareswaran K, Adamson R. Pump Position Impacts HeartMate II Left Ventricular Assist Device Thrombosis. ASAIO J. 2019 Mar/Apr;65(3):227-232. doi: 10.1097/MAT.0000000000000840. PMID 29952801
- [Derived] Thenappan T, Stulak JM, Agarwal R, Maltais S, Shah P, Eckman P, Emani S, Katz JN, Gregoric I, Keebler ME, Uriel N, Adler E, Chuang J, Farrar DJ, Sundareswaran KS, John R. Early intervention for lactate dehydrogenase elevation improves clinical outcomes in patients with the HeartMate II left ventricular assist device: Insights from the PREVENT study. J Heart Lung Transplant. 2018 Jan;37(1):25-32. doi: 10.1016/j.healun.2017.10.017. Epub 2017 Oct 24. PMID 29153636